CLINICAL TRIAL: NCT05104957
Title: Evaluation of the Kinesiology Taping Effectiveness in the Treatment of Lumbar Spine Pain in Subjects Under 30 Years of Age
Brief Title: Evaluation of the Kinesiology Taping Effectiveness in the Treatment of Lumbar Spine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II University in Biała Podlaska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PopeJohnPaulIIStateSchHigherE2
Record Dates: First submitted 2021-10-18; First posted 2021-11-03 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain; Young Adult; Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The study participants will be randomly qualified (allocated via a computer program) to the two groups: A - dynamic tape, B - sham (paper) tape
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Before commencing the tests, each participant was familiarized with their course, expressed their informed written consent for participation and random assignment to a specified tested group. The author of this paper had no influence on the categorization of the participants into individual treatment groups. During the studies, the physiotherapists performing the categorization were not informed about the results of the used treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic tape (Experimental): Experimental group will use a special dynamic tape on the lumbar extensor muscles
  Interventions: Other: Dynamic tape
- Paper tape (Sham Comparator): Control group will use a paper tape on the lumbar extensor muscles
  Interventions: Other: Sham tape

INTERVENTIONS:
Other: Dynamic tape — The experimental group will use a special dynamic patch made of cotton, coated with a hypoallergenic acrylic heat-activated adhesive arranged in sinusoidal-shaped layers. The tape will be applied using the muscle technique with a Y-shaped cut patch directly to the dried and non-greased skin. The application will be performed in a standing position, with the participant's lower extremities straight. The therapist will place the beginning of the tape (the base) on the participant's sacrum and then, asking them to bend 45 degrees forward, tape the tails of the tape along the spine on the extensor muscles of the lumbar region, without changing the tension of the tape, keeping the base in the initial position.
  Arms: Dynamic tape
Other: Sham tape — In the control group, a plain paper patch will be used to conduct the study, which, like the dynamic patch, will be applied using the same form of tape cutting and the same application technique. The entire method of applying the patch will also take place in the participant's standing position with forward bending. The paper patch will be placed at the levels from the L3 segment to the sacrum, along the spine on the lumbar extensor muscles.
  Arms: Paper tape

SUMMARY:
Lumbar spine pain syndromes are one of the most common pain conditions in our society.

The purpose of kinesiotaping is to normalize muscle function, improve blood and lymph flow, reduce pain, improve proprioception, promote tissue healing and restore normal tissue function. Today, this method is used in many fields of medicine. Its primary purpose is to support the musculoskeletal system by using various types of applications.

There is a lack of publications in the global literature on the effect of kinesiotaping of the external oblique muscles on lumbar spine pain. The main objective of this study is to evaluate the effectiveness of kinesiology taping in the treatment of lumbar spine pain in individuals under 30 years of age.

DETAILED DESCRIPTION:
Back pain occurs in people of all ages, regardless of their job. Both blue-collar and white-collar workers are exposed to strain and pain in the lumbar spine. The presence of pain is also promoted by low physical activity, poor motor habits, as well as stress.

There are numerous factors affecting the quality of life in patients with lower back pain. These include degree of pain, physical fitness, individual factors, degree of social support, and a potential for adapting forces to match constantly changing conditions.

The contemporary functional model of lumbar spinal muscles divides them into local stabilizers, single-joint global stabilizers, and multi-joint global stabilizers. The abdominal external oblique muscles are classified as global stabilizers. They generate force to control range of motion and allow limitation of that range (eccentric control), and functionally control rotation in all movements, regardless of the load acting on the spine.

The main objective of this study is to evaluate the effectiveness of kinesiology taping in the treatment of lumbar spine pain in individuals under 30 years of age.

ELIGIBILITY:
Inclusion Criteria:

* participants' age between 18 and 30,
* the presence of pain in the lumbar region of the spine,
* participants who have not been using non-steroidal anti-inflammatory drugs (NSAIDs) for at least one week prior to study entry,
* no contraindications to the use of dynamic kinesiology taping patches,
* informed, written consent to participate in the study.

Exclusion Criteria:

* status of the post lumbar spine surgery,
* subjects who have had a spinal injury within 6 months prior to the start of the study,
* neoplastic diseases,
* congenital structural pathologies of the spine,
* allergy to the adhesive substance of kinesiology taping or paper patch,
* being a physiotherapy student.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of pain (VAS) | Visual analogue pain scale (VAS) will be carried out before the start of the therapy.
  Visual analogue scale of pain (VAS) evaluates intensity of pain in the scale from 0 to 10. Maximum score means the highest level of pain.
Visual analogue scale of pain (VAS) | Visual analogue pain scale (VAS) will be carried out 4 days of therapy, immediately after its completion.
  Visual analogue scale of pain (VAS) evaluates intensity of pain in the scale from 0 to 10. Maximum score means the highest level of pain.
Visual analogue scale of pain (VAS) | Visual analogue pain scale (VAS) will be carried out four weeks after the end of the treatment.
  Visual analogue scale of pain (VAS) evaluates intensity of pain in the scale from 0 to 10. Maximum score means the highest level of pain.

SECONDARY OUTCOMES:
Modified Laitinen's pain questionnaire | Modified Laitinen's pain questionnaire will be carried out three times (before the start of the therapy, after 4 days of therapy, immediately after its completion and four weeks after the end of the treatment
  The Laitinen questionnaire takes into account four indicators evaluated in a scale of 0 to 4: the intensity of pain, the frequency of its occurrence, the use of analgesic medications and limitation of the participant's motor activity. A research participant could be granted from 0 to 16 points, the maximum score meaning the highest level of pain.
Oswestry Disability Index | Oswestry Disability Index will be carried out three times (before the start of the therapy, after 4 days of therapy, immediately after its completion and four weeks after the end of the treatment
  Oswestry Disability Index takes into account ten indicators evaluated in a scale of 0 to 5. A research participant could be granted from 0 to 50 points, the minimum score meaning the highest level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Zaworski, Ph.D., Study Chair — John Paul II University in Biała Podlaska
Locations (2):
- Poland (2):
  - Pope John Paul II State School Of Higher Education in Biała Podlaska, Biała Podlaska
  - Laboratory of Pope John Paul II State School Of Higher Education in Biala Podlaska, Biała Podlaska

IPD SHARING:
Plan to Share IPD: No